CLINICAL TRIAL: NCT04627090
Title: Langerhans Cell Histiocytosis in Adults: a Collaborative, Prospective-retrospective, Observational GIMEMA Study
Brief Title: LCH in Adults: a Collaborative, Prospective-retrospective, Observational Study
Status: Recruiting | Type: Observational
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: RD0120
Record Dates: First submitted 2020-11-02; First posted 2020-11-13 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Langerhans Cell Histiocytosis
MeSH Terms: conditions — Histiocytosis, Langerhans-Cell | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LCH Patients: Adult patients with LCH, diagnosed starting from January 2001
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Diagnostic and therapeutic data of adult patients with LCH, collected from clinical and laboratory evaluations, carried out during clinical practice.

SUMMARY:
This is a multicenter, retrospective and prospective, observational, no profit study including adult patients with LCH, diagnosed starting from January 2001 to two years after the first enrolled patient. Each patient will be followed up to one year after the last enrolled patient. Each patient will be followed up to one year after the last enrolled patient.This study plans to collect clinical information at the time of diagnosis and at various follow-ups to evaluate the efficacy of first-line therapies. Diagnostic and therapeutic data will be collected from routine clinical evaluations and laboratory and instrumental investigations carried out during clinical practice

DETAILED DESCRIPTION:
This is a multicenter, retrospective and prospective, observational, no profit study including adult patients with LCH, diagnosed starting from January 2001 to two years after the first enrolled patient. Data from patients, diagnosed from January 2001 to the date of patient enrolment, is considered retrospective, while data collected after patient enrolment, and up to two years after the first enrolled patient, is considered prospective. At least one year of follow-up is expected for each patient. Each patient will be followed up to one year after the last enrolled patient. This study plans to collect clinical information at the time of diagnosis and at various follow-ups to evaluate the efficacy of first-line therapies. Diagnostic and therapeutic data will be collected from routine clinical evaluations and laboratory and instrumental investigations carried out during clinical practice. A sub-cohort of patients with available biological data on somatic mutations of the RAF-MEK-ERK genes will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed histological and immunohistochemical diagnosis of LCH (CD1a+, S-100+, CD207+), from January 2001 up to two years after the first enrolled patient. Patients with isolated vertebra plana, not related to a malignancy, and without a soft tissue component, are included without a histological and immunohistochemical diagnosis;
* Age ≥18 years at the time of definitive diagnosis;
* Signed, written informed consent, according to ICH/EU/GCP, and national, local laws.

Exclusion Criteria:

* Age ≥18 years and presumptive diagnosis of LCH, or definitive diagnosis of non-Langerhans Histiocytosis (Juvenile xantogranuloma, Rosai-Dorfman disease, Erdheim-Chester disease, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients with LCH, diagnosed starting from January 2001 to two years after the first enrolled patient.
Sampling Method: Non-Probability Sample
Enrollment: 186 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Evaluation of efficacy of first-line therapies | up to 3 months
  Number of patients who achive complete/intermediate response

CONTACTS AND LOCATIONS:
Locations (8):
- Italy (8):
  - Ao Brotzu, Presidio Ospedaliero A. Businco - Cagliari - Sc Ematologia E Ctmo, Cagliari
  - Ctc U.O Di Ematologia Con Trapianto Di Midollo Osseo - Catania, Catania
  - Fondazione Irccs "Istituto Nazionale Tumori" - Milano - Sc Ematologia, Milan
  - Ao Regionale S. Carlo - Potenza - Sic Ematologia, Potenza
  - Fondazione Policlinico Universitario Agostino Gemelli Irccs, Roma
  - Università Degli Studi Di Roma "Sapienza" - Dipartimento Di Medicina Traslazionale E Di Precisione - U.O.C. Ematologia, Roma
  - Aou "San Giovanni Di Dio E Ruggi D'Aragona" - Salerno - Uoc Ematologia E Trapianti Di Cellule Staminali Emopoietiche, Salerno
  - Aou Di Sassari - Cliniche Universitarie - Stabilimento Cliniche Di San Pietro - Uoc Ematologia, Sassari